CLINICAL TRIAL: NCT03469310
Title: Minimizing Narcotic Analgesics After Thyroid or Parathyroid Surgery
Brief Title: Minimizing Narcotic Analgesics After Endocrine Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Minerva A Romero Arenas (Other)
Responsible Party: Sponsor-Investigator, Minerva A Romero Arenas, Principal Investigator, DHR Health Institute for Research and Development
Organization: DHR Health Institute for Research and Development (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1177315
Record Dates: First submitted 2018-03-07; First posted 2018-03-19 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Thyroid Cancer; Thyroid Nodule; Thyroid Neoplasms; Thyroid Goitre; Thyroid Diseases; Parathyroid Diseases; Parathyroid Adenoma; Parathyroid Hyperplasia
Keywords: endocrine surgery; opioid addiction; pain management; analgesia
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Nodule; Goiter; Thyroid Diseases; Parathyroid Diseases; Parathyroid Neoplasms; Opioid-Related Disorders; Agnosia | interventions — Acetaminophen; Capsules; acetaminophen, codeine drug combination; Tramadol

STUDY DESIGN:
Intervention Model Description: option 1: Tylenol (also known as acetaminophen) with tramadol if needed, or option 2: Tylenol #3 as needed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acetaminophen (Experimental): Tylenol (also known as acetaminophen) 1000mg every 6 hours for 3 days and tramadol 50 mg every 6 hours as needed for moderate to severe pain
  Interventions: Drug: Acetaminophen 500Mg Cap; Drug: Tramadol
- Codeine Acetaminophen (Active Comparator): Tylenol #3 (codeine-acetaminophen) 1 tab every 4 hours or 2 tabs every 6 hours as needed for pain
  Interventions: Drug: Tylenol #3 Oral Tablet

INTERVENTIONS:
Drug: Acetaminophen 500Mg Cap — non-narcotic medication first with narcotic as second choice
  Other Names: Tylenol
  Arms: Acetaminophen
Drug: Tylenol #3 Oral Tablet — Narcotic medication first
  Other Names: codeine-acetaminophen
  Arms: Codeine Acetaminophen
Drug: Tramadol — non-narcotic medication first with narcotic as second choice
  Arms: Acetaminophen

SUMMARY:
This research is being done to better understand and test if the investigators can minimize narcotic medication for controlling pain after thyroid or parathyroid surgery. This research will be performed at Doctors Hospital At Renaissance in the investigators clinic and the perioperative area.

Participants will be randomly chosen to receive one of two options for pain management that the investigators are already using in the care of patients after surgery. One option includes a narcotic medication and one option includes a non-narcotic and a narcotic as needed.

Participants will be asked to complete a form about the level of pain and how much pain medication was needed after surgery in the hospital and while at home. Participants will not have to do any additional visits to participate in this study. The investigators will obtain the research materials at the same time as the usual care visits around the participants' surgery.

DETAILED DESCRIPTION:
A study team member will give the participant a copy of the informed consent form to read. Participants will have a chance to ask questions about the study before agreeing to participate. If participants agree, they will be randomly chosen to receive one of two options for pain management that the investigators are already using in the care of patients (option 1: Tylenol (also known as acetaminophen) with tramadol if needed, or option 2: Tylenol #3 as needed) after surgery.

Participants will be asked to complete a form about the level of pain and how much pain medication was needed after surgery in the hospital and while at home. Participants will come to the GME General Surgery Center approximately one week after surgery for a post-operative visit so that the investigators can see how much pain medication was used and how much pain the participant had in the first few days after surgery.

Participants will not have to do any additional visits to participate in this study. The investigators will obtain the research materials at the same time as the usual care visits around the participants' surgery. It should take approximately 2 minutes each day to complete.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients 18 years of age or older,
2. Who are undergoing thyroid or parathyroid surgery at DHR by an Endocrine Surgery faculty member,
3. Provide informed consent to participate in the study in English or Spanish,
4. Patients will be included if they are discharged the same day or on postoperative day 1,
5. Patients who undergo central lymphadenectomy will be included,
6. Patients who undergo two operations within a 2-week period (for example a thyroid lobectomy followed by subsequent completion thyroidectomy) will only have the postoperative narcotic requirements following the initial operation included for the study analysis.
7. Patients who have a complication, such as seroma or hematoma, requiring return to the operating room within 48 hours will be included in the study for the initial operation only.

Exclusion Criteria:

1. Patients who undergo lateral neck lymph node dissection will be excluded from the study due to the extent of the operation requiring a different analgesic regimen;
2. Patients allergic to any of the study drugs will be ineligible;
3. Patients who undergo two operations within a 2-week period (for example a thyroid lobectomy followed by subsequent completion thyroidectomy) will only have the initial operation included for the study analysis.
4. Patients with a formal diagnosis of hepatic failure will be ineligible
5. Patients with any diagnosis of chronic pain requiring treatment with ongoing narcotic regimen will be ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2019-12-21 (Actual); Study Completion 2020-10-02 (Actual)

PRIMARY OUTCOMES:
Staged narcotic analgesic regimen is non-inferior to narcotics in controlling pain | Patient will report pain score up to two weeks after surgery
  Patient pain scores will be logged using Wong-Baker FACES pain rating scale (range 0-10) and scores will be assessed for differences between the study arms

SECONDARY OUTCOMES:
Is there a difference in the duration of postoperative pain requiring medication | Patient will report medication requirements up to two weeks after surgery
  The number of days after surgery that participants required pain medications will be counted and assessed for difference between the study arms
Is there a difference in the medication requirement | Patient will report medication requirements up to two weeks after surgery
  The type and quantity of pain medications used after surgery will be counted and assessed for difference between the study arms
Staged regimen cross over to narcotic | Patient will report medication requirements up to two weeks after surgery
  The type and quantity of pain medications used after surgery will be counted and number of patients requiring cross over will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Minerva A Romero Arenas, MD, MPH, Principal Investigator — GME General Surgery; Samuel K Snyder, MD, Principal Investigator — GME General Surgery; Henry A Reinhart, MD, Principal Investigator — GME General Surgery
Locations (1):
- GME General Surgery Clinic, Edinburg, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified information only will be made available to interested researchers.
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Background] Rudd RA, Seth P, David F, Scholl L. Increases in Drug and Opioid-Involved Overdose Deaths - United States, 2010-2015. MMWR Morb Mortal Wkly Rep. 2016 Dec 30;65(50-51):1445-1452. doi: 10.15585/mmwr.mm655051e1. PMID 28033313
- [Background] Waljee JF, Li L, Brummett CM, Englesbe MJ. Iatrogenic Opioid Dependence in the United States: Are Surgeons the Gatekeepers? Ann Surg. 2017 Apr;265(4):728-730. doi: 10.1097/SLA.0000000000001904. No abstract available. PMID 27429023
- [Background] Jiang X, Orton M, Feng R, Hossain E, Malhotra NR, Zager EL, Liu R. Chronic Opioid Usage in Surgical Patients in a Large Academic Center. Ann Surg. 2017 Apr;265(4):722-727. doi: 10.1097/SLA.0000000000001780. PMID 27163960
- [Background] Dowell D, Haegerich TM, Chou R. CDC Guideline for Prescribing Opioids for Chronic Pain - United States, 2016. MMWR Recomm Rep. 2016 Mar 18;65(1):1-49. doi: 10.15585/mmwr.rr6501e1. PMID 26987082
- [Background] Scully RE, Schoenfeld AJ, Jiang W, Lipsitz S, Chaudhary MA, Learn PA, Koehlmoos T, Haider AH, Nguyen LL. Defining Optimal Length of Opioid Pain Medication Prescription After Common Surgical Procedures. JAMA Surg. 2018 Jan 1;153(1):37-43. doi: 10.1001/jamasurg.2017.3132. PMID 28973092
- [Background] Rogers SO Jr. Addressing Variability in Opioid Prescribing. JAMA Surg. 2018 Jan 1;153(1):43. doi: 10.1001/jamasurg.2017.3166. No abstract available. PMID 28973361